CLINICAL TRIAL: NCT01040104
Title: Pilot Study of Prospective Clinical Trials on Skin Wound Healing in Young and Aged Individuals
Brief Title: Prospective Clinical Trials on Skin Wound Healing in Young and Aged Individuals
Acronym: RESOLVE
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, David Lumenta, MD, Dr, Medical University of Vienna
Other Study IDs: FP7-202047.WP.2.1-2.2-2.4; MUW-EK-Nr_015/2009 (Other: MUVienna)
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Age; Cicatrix, Hypertrophic; Fibrosis; Diabetes Mellitus
Keywords: wound healing; hypertrophic scar; skin transplantation; diabetes mellitus
MeSH Terms: conditions — Cicatrix, Hypertrophic; Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsy Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Regular wound healing, young: Regular skin repair, controlled wound healing conditions in young individuals
  Interventions: Other: Skin sample; Other: Blood taking
- Regular wound healing, aged: Regular skin repair, controlled wound healing conditions in aged individuals
  Interventions: Other: Skin sample; Other: Blood taking
- Hypertrophic scarring, young: Skin repair with and without hypertrophic scarring in young individuals
  Interventions: Other: Skin biopsy; Other: Blood taking
- Hypertrophic scarring, aged: Skin repair with and without hypertrophic scarring in aged individuals
  Interventions: Other: Skin biopsy; Other: Blood taking
- Non-diabetic, young: Skin repair in non-diabetic young individuals
  Interventions: Other: Skin biopsy; Other: Blood taking
- Non-diabetic, aged: Skin repair in non-diabetic aged individuals
  Interventions: Other: Skin biopsy; Other: Blood taking
- Diabetic, young: Skin repair in young diabetic individuals
  Interventions: Other: Skin biopsy; Other: Blood taking
- Diabetic, aged: Skin repair in aged diabetic individuals
  Interventions: Other: Skin biopsy; Other: Blood taking

INTERVENTIONS:
Other: Skin sample — Taken from regularly discarded tissue during routine operation
  Groups: Regular wound healing, aged; Regular wound healing, young
Other: Skin biopsy — Skin biopsy from regions exhibiting normal and/or hypertrophic scarring at day 0 and day 90
  Groups: Hypertrophic scarring, aged; Hypertrophic scarring, young
Other: Skin biopsy — Biopsy from skin graft harvest site during routine operation on day 0 and follow-up on day 90
  Groups: Diabetic, aged; Diabetic, young; Non-diabetic, aged; Non-diabetic, young
Other: Blood taking — Blood taking on day 0
Other: Blood taking — Blood taking on day 90
  Groups: Diabetic, aged; Diabetic, young; Hypertrophic scarring, aged; Hypertrophic scarring, young; Non-diabetic, aged; Non-diabetic, young

SUMMARY:
Regular wound healing follows a well-ordered sequence of overlapping phases: inflammation, proliferation, maturation and remodelling.

In the young, damage to an organ mostly triggers fully regenerative mechanisms called "primary" wound healing. Repeated damage in young individuals may cause "secondary" wound healing eg. scar formation reflecting a rescue program, in which reorganisation has failed.

Organ failure in the ageing organism is characterized by a progressive loss of its capability to achieve an orderly reactivation of organ repair, and results in a combination of chronic inflammation and fibroproliferative, non-regenerative repair affecting several organs, including lung, liver and skin.

RESOLVE's objective is to identify, characterize, and validate molecular targets responsible for shifting primary organ repair towards fibroproliferative wound healing as a result of an age-dependent loss of regulatory control.

The structured approach is based on

* different forms of wound healing,
* different human diseases and
* different genetic backgrounds,

aiming to provide future diagnostic tools in various organs, to create transgenic animal test systems, and to identify molecular targets involved in fibroproliferative wound healing.

DETAILED DESCRIPTION:
Cutaneous scars are frequently encountered conditions. The process of wound repair, however, is complicated, and various factors contribute to different types of scarring (eg. hypertrophic, atrophic).

WP 2.1: Regular skin repair

In elective plastic surgery most excised operative skin specimens are usually discarded, and represent an excellent opportunity of harvesting skin biopsies without additional invasive measures. This work package analyzes skin samples of individuals after elective plastic surgery with normal wound healing serving as control group.

WP 2.2: Skin repair with and without hypertrophic scar formation

A classic example of fibroproliferative repair in the skin is hypertrophic scarring classified as a dermal skin lesion, which is raised above skin level, stays within the confines of the initial wound and increases in size by pushing out the margins of the scar without invading the surrounding normal tissue.

Hypertrophic scarring is a condition commonly observed after burns and in regions of prolonged wound healing (>21 days). The underlying pathology of hypertrophic scarring, however, is poorly understood. Hypertrophic scars can be managed conservatively, and only require surgical intervention under special circumstances.

This work package analyzes the clinical and molecular response to a standard treatment regimen in skin regions with and without hypertrophic scars after skin injuries.

WP 2.4: Wound healing in normal and diabetic individuals

Diabetes mellitus is a known factor to cause impaired wound healing. Due to microangiopathic, macroangiopathic and other conditions resulting from atherosclerosis and peripheral neuropathy wound healing in diabetic individuals is usually delayed (hypotrophic, atrophic) and often complicated by immunosuppression and superinfections. The rising prevalence of diabetes mellitus in the elderly population makes it necessary to understand its related processes in relevant clinical wound models.

Split-thickness skin-grafting is a commonly applied technique in plastic surgery, and donor sites of previously uninjured skin regions spontaneously heal within two weeks, representing an ideal condition to monitor clinical and molecular changes in diseased vs. non-diseased states.

This work package analyzes skin repair in donor sites of split-thickness skin grafts in non-diabetic and diabetic individuals.

ELIGIBILITY:
WP2.1

Inclusion Criteria:

* age 18-45 and 55-85 years, respectively

Exclusion Criteria:

* past medical history of hypertrophic scarring or keloid disease
* cardiac disease adversely affecting peripheral blood flow
* active neoplastic disease
* immunosuppressive condition, congenital or acquired
* anemia
* autoimmune disorder
* acute or chronic renal failure
* liver cirrhosis or active hepatitis
* active substance-abuse disorder
* severe underweight (body mass index <16)
* endocrinological disorder
* pregnancy or lactation for women of child-bearing age

WP2.2

Inclusion Criteria:

* age 18-45 and 55-85 years, respectively
* normal and/or hypertrophic scars
* Baux score <100

Exclusion Criteria:

* sepsis
* electrical and/or chemical burn
* clinically significant wound infection in areas of planned biopsies
* cardiac disease adversely affecting peripheral blood flow
* active neoplastic disease
* immunosuppressive condition, congenital or acquired
* autoimmune disorder
* acute or chronic renal failure
* liver cirrhosis or active hepatitis
* active substance-abuse disorder
* severe underweight (body mass index <16)
* endocrinological disorder
* pregnancy or lactation for women of child-bearing age

WP 2.4

Inclusion Criteria:

* age 18-45 and 55-85 years, respectively

Exclusion Criteria:

* cardiac disease adversely affecting peripheral blood flow
* active neoplastic disease
* immunosuppressive condition, congenital or acquired
* anemia
* autoimmune disorder
* acute or chronic renal failure
* liver cirrhosis or active hepatitis
* substance-abuse disorder
* severe underweight (body mass index <16)
* thyroid function disorder
* pregnancy or lactation for women of child-bearing age

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: WP 2.1 Individuals due for planned elective plastic surgery with regular wound healing
  WP 2.2 Individuals, who suffered from burns, trauma or having undergone any type of previous surgery with and without hypertrophic scar formation
  WP 2.4 Individuals, who require split-thickness skin grafting for skin defects with or without diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Time to wound healing / Scar maturation | day14, day90, day180

CONTACTS AND LOCATIONS:
Overall Officials: Lars P Kamolz, MD, MSc, Principal Investigator — MUW
Locations (1):
- Division of Plastic and Reconstructive Surgery, Department of Surgery, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Gangemi EN, Gregori D, Berchialla P, Zingarelli E, Cairo M, Bollero D, Ganem J, Capocelli R, Cuccuru F, Cassano P, Risso D, Stella M. Epidemiology and risk factors for pathologic scarring after burn wounds. Arch Facial Plast Surg. 2008 Mar-Apr;10(2):93-102. doi: 10.1001/archfaci.10.2.93. PMID 18347236
- [Background] Izadi K, Ganchi P. Chronic wounds. Clin Plast Surg. 2005 Apr;32(2):209-22. doi: 10.1016/j.cps.2004.11.011. PMID 15814118
- [Background] Blakytny R, Jude E. The molecular biology of chronic wounds and delayed healing in diabetes. Diabet Med. 2006 Jun;23(6):594-608. doi: 10.1111/j.1464-5491.2006.01773.x. PMID 16759300
- [Background] Komesu MC, Tanga MB, Buttros KR, Nakao C. Effects of acute diabetes on rat cutaneous wound healing. Pathophysiology. 2004 Oct;11(2):63-67. doi: 10.1016/j.pathophys.2004.02.002. PMID 15364115
- [Background] Niessen FB, Spauwen PH, Schalkwijk J, Kon M. On the nature of hypertrophic scars and keloids: a review. Plast Reconstr Surg. 1999 Oct;104(5):1435-58. doi: 10.1097/00006534-199910000-00031. No abstract available. PMID 10513931
- [Background] Rockwell WB, Cohen IK, Ehrlich HP. Keloids and hypertrophic scars: a comprehensive review. Plast Reconstr Surg. 1989 Nov;84(5):827-37. doi: 10.1097/00006534-198911000-00021. No abstract available. PMID 2682703
- [Background] Gottrup F, Agren MS, Karlsmark T. Models for use in wound healing research: a survey focusing on in vitro and in vivo adult soft tissue. Wound Repair Regen. 2000 Mar-Apr;8(2):83-96. doi: 10.1046/j.1524-475x.2000.00083.x. PMID 10810034
- [Background] Ashcroft GS, Mills SJ, Ashworth JJ. Ageing and wound healing. Biogerontology. 2002;3(6):337-45. doi: 10.1023/a:1021399228395. PMID 12510172
- [Background] Gosain A, DiPietro LA. Aging and wound healing. World J Surg. 2004 Mar;28(3):321-6. doi: 10.1007/s00268-003-7397-6. Epub 2004 Feb 17. PMID 14961191
- [Background] Crooks A. How does ageing affect the wound healing process? J Wound Care. 2005 May;14(5):222-3. doi: 10.12968/jowc.2005.14.5.26777. PMID 15909438
- [Background] Deitch EA, Wheelahan TM, Rose MP, Clothier J, Cotter J. Hypertrophic burn scars: analysis of variables. J Trauma. 1983 Oct;23(10):895-8. PMID 6632013
- [Background] Bombaro KM, Engrav LH, Carrougher GJ, Wiechman SA, Faucher L, Costa BA, Heimbach DM, Rivara FP, Honari S. What is the prevalence of hypertrophic scarring following burns? Burns. 2003 Jun;29(4):299-302. doi: 10.1016/s0305-4179(03)00067-6. PMID 12781605
- [Background] Oliveira GV, Chinkes D, Mitchell C, Oliveras G, Hawkins HK, Herndon DN. Objective assessment of burn scar vascularity, erythema, pliability, thickness, and planimetry. Dermatol Surg. 2005 Jan;31(1):48-58. doi: 10.1111/j.1524-4725.2005.31004. PMID 15720096
- [Background] Mustoe TA, Cooter RD, Gold MH, Hobbs FD, Ramelet AA, Shakespeare PG, Stella M, Teot L, Wood FM, Ziegler UE; International Advisory Panel on Scar Management. International clinical recommendations on scar management. Plast Reconstr Surg. 2002 Aug;110(2):560-71. doi: 10.1097/00006534-200208000-00031. PMID 12142678
- See also: Ethics Committee of the Medical University of Vienna and the Vienna General Hospital — http://www.meduniwien.ac.at/ethik/index.htm